CLINICAL TRIAL: NCT05465759
Title: Frequency of SARS COV-2 Infection Among Malignant Patients at South Egypt Cancer Institute
Brief Title: Frequency of SARS COVID-19 Infection Among Malignant Patients at South Egypt Cancer Institute
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Agamy, Principal investigator, Assiut University
Other Study IDs: COVID-19 in cancer patients
Record Dates: First submitted 2022-07-13; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: disease — Frequency of SARS COV-2 infection among malignant patients at south Egypt Cancer institute.

SUMMARY:
Assessment the frequency of SARS COV-2 infection among malignant patients at south Egypt Cancer institute

DETAILED DESCRIPTION:
Coronavirus disease (COVID-19) is an infectious disease caused by the SARS-CoV-2 virus Most people infected with the virus will experience mild to moderate respiratory illness and recover without requiring special treatment. However, some will become seriously ill and require medical attention. Older people and those with underlying medical conditions like cardiovascular disease, diabetes, chronic respiratory disease, or cancer are more likely to develop serious illness. Anyone can get sick with COVID-19 and become seriously ill or die at any age Cancer is one of the most common examples of immunocompromised states

ELIGIBILITY:
Inclusion Criteria:

* Malignant patients.
* PCR positive for covid-19

Exclusion Criteria:

* PCR negative for covid-19

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients at south Egypt cancer institute
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
calculate the frequency of SARS-CoV-2 infection among patients with malignant data collection during the study period | 1 year
  To calculate the rate of SARS-CoV-2 infection among patients with malignant data collection within covid-19 pandemic either retrospective or prospective.
  Data will include :
  patient demography such as Age,sex,smoking status,cancer type cancer treatment (patient on chemotherapy or radiotherapy if available), symptoms, signs and laboratory parameters of COVID -19. outcome including hospitalization or ICU admission and mortality rate will be recorded